CLINICAL TRIAL: NCT03714828
Title: A Single Arm Phase 2 Study of Talimogene Laherparepvec in Patients With Cutaneous Squamous Cell Cancer
Brief Title: Study of TVEC in Patients With Cutaneous Squamous Cell Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Arizona (Other)
Collaborators: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1807738975; 29088 (Other: University of Arizona Cancer Center)
Record Dates: First submitted 2018-10-08; First posted 2018-10-22 (Actual); Results first posted 2024-10-09 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-10

CONDITIONS: Squamous Cell Carcinoma; Skin Cancer; Keratoacanthoma; Cutaneous Tumor; Skin Cancer, Squamous Cell; Lesion Skin
Keywords: Skin cancer; Squamous cell; Squamous Cell Carcinoma; Skin lesion; Keratoacanthoma; talimogene laherparepvec
MeSH Terms: conditions — Carcinoma, Squamous Cell; Skin Neoplasms; Keratoacanthoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Treatment (talimogene laherparepvec) (Experimental): The subject participation period will be approximately 48 weeks. This will include a screening visit, 4 injection visits and 5 follow up visits. Total length of study/patient is 8.5 to 10.5 months. TVEC will be administered by injection with a needle directly into one or more tumors.
  Interventions: Drug: Injection of TVEC into target lesions - week 1-2; Drug: Injection of TVEC into target lesions 3wks after 1st injection; Drug: Injection of TVEC into target lesions 2wks after 2nd injection; Drug: Injection of TVEC into target lesions 2wks after 3rd injection

INTERVENTIONS:
Drug: Injection of TVEC into target lesions - week 1-2 — Target lesions are identified and documented with measurements and photographs. Photographs will be taken with regional and close up view of the anatomical area and lesion.
  Inject 0.5ml - 4ml (based on lesion size - section 7.1, Table 5) Talimogene laherparepvec at nominal concentration of 106 plaque forming units (PFU)/mL with approximately 1.15 mL in a 2 mL vial for the initial dose. This will be administered intralesionally to 1-3 cSCC lesions per anatomical site with a maximum of 5 injectable lesions per patient.
Drug: Injection of TVEC into target lesions 3wks after 1st injection — Target lesions are identified and documented with measurements and photographs. Photographs will be taken with global and close up view of the anatomical area and lesion.
  Inject 0.5ml - 4ml (based on lesion size) and number of lesions selected. Talimogene laherparepvec at nominal concentration of 108 PFU/mL with approximately 1.15 mL in a 2 mL vial for the second and subsequent doses.
Drug: Injection of TVEC into target lesions 2wks after 2nd injection — Target lesions are identified and documented with measurements and photographs. Photographs will be taken with global and close up view of the anatomical area and lesion.
  Inject 0.5ml - 4ml (based on lesion size) and number of lesions selected.Talimogene laherparepvec at nominal concentration of 108 PFU/mL with approximately 1.15 mL in a 2 mL vial for the subsequent doses.
Drug: Injection of TVEC into target lesions 2wks after 3rd injection — Target lesions are identified and documented with measurements and photographs. Photographs will be taken with global and close up view of the anatomical area and lesion.
  Inject 0.5ml - 4ml (based on lesion size) and number of lesions selected. Talimogene laherparepvec at nominal concentration of 108 PFU/mL with approximately 1.15 mL in a 2 mL vial for the subsequent doses.

SUMMARY:
This is single arm Phase 2, single center study of talimogene laherparepvec (TVEC) to treat low risk cutaneous squamous cell carcinomas (cSCC).

DETAILED DESCRIPTION:
The purpose of this study is to assess the effect of Talimogene laherparepvec (TVEC) in patients diagnosed with lower risk cSCC in need of alternative therapeutic approaches.

Immune recognition and cytotoxic responses play an important role in the pathogenesis and progression of cutaneous squamous cell carcinoma (cSCC). TVEC is an HSV-1 oncolytic immunological agent FDA approved for the local treatment of unresectable recurrent melanoma. It is proposed that T-VEC directly destroys cancer cells and induces production of GM-CSF to enhance systemic antitumor immune priming. This proposed mechanism of action supports the novel approach to implement TVEC in the management of cSCC. Particularly, in patients with increased burden of primary tumors.

The study subjects enrolled in the study were Immunocompetent, > 18 years of age, and diagnosed with at least one histologically confirmed primary low-risk cSCC according to the Brigham and Women staging system. Unresectable lesions or patients unable/unwilling to undergo standard of care treatment were eligible to participate. Study lesions included target lesions injected (TLIs) and target non-injected lesions (TNILs). TNILs were selected to evaluate for abscopal effect when feasible. The TLIs were treated according to TVEC FDA approved protocol and followed for 1yr after the 1st injection. The primary endpoint of the study was to evaluate the overall response rate, defined as the proportion of subjects who achieved complete response and partial response in the TLIs. Safety and adverse effect profile (AEs), duration of response, time to response, durable response rate, and time to progression, were the some of the secondary endpoints included.

ELIGIBILITY:
Inclusion Criteria:

1. Able to give informed consent in English or Spanish
2. Age > 18
3. Have at least one >0.5 cm to <5.0 cm, histologically confirmed low risk cutaneous SCC (including kerathoacanthomas)

   * Size >0.5 cm on trunk or extremities (excluding face, neck feet, nail units, and ankles)
   * Clinically consistent with primary tumors.
   * Lesion considered unresectable (as defined in Section 1.2)
   * Recurrent lesions will be considered eligible if additional inclusion criteria are met.
   * No immunosuppression
   * Not a site of previous radiation therapy or chronic significant inflammation
   * Fast growing lesions (doubling in size over a 4 week period of time) will be included if they are clinically suggestive of cSCC of the keratoacanthoma type.
   * Well or moderately differentiated tumor as confirmed by skin biopsy
   * Depth less than 2 mm (for non KA type cSCC )
   * No perineural or vascular involvement in preliminary biopsy.
4. Partial biopsy of squamous cell skin cancer identified as a target lesion(s) to determine the histological differentiation of the tumor or other adverse histological features
5. In patients with multiple lesions, up to 3 lesions in a similar anatomical site, (trunk, limbs etc) that is at least 10 cm apart can be selected.
6. Maximum of 5 lesions per patient can be selected for treatment
7. Adequate organ function determined within 28 days prior to enrollment, defined as follows:
8. Hematology:

   * Absolute neutrophil count ≥ 1500/mm3 (1.5x109/L)
   * Platelet count ≥ 75,000/mm3 (7.5x109/L)
   * Hemoglobin ≥ 8 g/dL (without need for hematopoietic growth factor or transfusion support)
9. Renal

   • Serum creatinine ≤ 1.5 x upper limit of normal (ULN), OR 24-hour creatinine clearance ≥ 60 mL/min for subject with creatinine levels > 1.5 x ULN. (Note: Creatinine clearance need not be determined if the baseline serum creatinine is within normal limits. Creatinine clearance should be determined per institutional standard)
10. Hepatic

    * Serum bilirubin ≤ 1.5 x ULN
    * Aspartate aminotransferase (AST) ≤ 2.5 x ULN 23 | Page Version 6-26-2018
    * Alanine aminotransferase (ALT) ≤ 2.5 x ULN
11. Coagulation

    * International normalization ratio (INR) or prothrombin time (PT) ≤ 1.5 x ULN, unless the subject is receiving anticoagulant therapy, in which case PT and partial thromboplastin time (PTT)/ activated PTT (aPTT) must be within therapeutic range of intended use of anticoagulants.
    * PTT or aPTT ≤ 1.5 x ULN unless the subject is receiving anticoagulant therapy as long as PT and PTT/aPTT is within therapeutic range of intended use of anticoagulants.
12. Female subject of childbearing potential should have a negative urine or serum pregnancy test within 72 hours prior to enrollment. If urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.

Exclusion Criteria:

1. Any patient with diagnosis of invasive cancer in the last 3 years with the exception of stage I and II melanoma, cutaneous BCC and SCCs will be excluded.
2. Subjects on acitretin, capecitabine, topical chemotherapies or treatments.
3. History or evidence of symptomatic autoimmune disease (eg, pneumonitis, glomerulonephritis, vasculitis, or other), or history of active autoimmune disease that has required systemic treatment (ie, use of corticosteroids, immunosuppressive drugs or biological agents used for treatment of autoimmune diseases) in past 2 months prior to enrollment. Replacement therapy (eg, thyroxine for hypothyroidism, insulin for diabetes or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency) is not considered a form of systemic treatment for autoimmune disease.
4. Evidence of clinically significant immunosuppression such as the following:

   * Primary immunodeficiency state such as Severe Combined Immuno deficiency Disease
   * Acquired immunodeficiency syndrome
   * Concurrent opportunistic infection
   * Receiving systemic immunosuppressive therapy (> 2 weeks) including oral steroid doses > 10 mg/day of prednisone or equivalent within 2 months prior to enrollment.
5. Active herpetic skin lesions or prior complications of herpetic infection (e.g., herpetic keratitis or encephalitis).
6. Requires intermittent or chronic systemic (intravenous or oral) treatment with an antiherpetic drug (e.g., acyclovir), other than intermittent topical use.
7. Previous treatment with talimogene laherparepvec or any other oncolytic virus
8. Prior therapy with tumor vaccine
9. Received live vaccine within 28 days prior to enrollment. 24 | Page Version 6-26-2018
10. Currently receiving treatment with another investigational device or drug study, or < 28 days since ending treatment with another investigational device or drug study(s)
11. Other investigational procedures while participating in this study are excluded.
12. Known to have acute or chronic active hepatitis B infection
13. Known to have acute or chronic active hepatitis C infection
14. History of other malignancy within the past 3 years with the following exceptions:

    * adequately treated mucosa associated lymphoid tissue (MALT) tumor
    * malignancy treated with curative intent and with no known active disease present for ≥ 3 years before enrollment and felt to be at low risk for recurrence by the treating physician
    * adequately treated non-melanoma skin cancer, lentigo maligna, stage I or II cutaneous melanoma, without evidence of disease.
    * adequately treated cervical carcinoma in situ without evidence of disease
    * adequately treated breast ductal carcinoma in situ without evidence of disease
    * prostatic intraepithelial neoplasia without evidence of prostate cancer
    * adequately treated urothelial papillary noninvasive carcinoma or carcinoma in situ
15. Subject has known sensitivity to talimogene laherparepvec or any of its components to be administered during dosing.
16. Female subject is pregnant or breast-feeding, or planning to become pregnant during study treatment and through 3 months after the last dose of talimogene laherparepvec
17. Female subject of childbearing potential who is unwilling to use acceptable method(s) of effective contraception during study treatment and through 3 months after the last dose of talimogene laherparepvec. (Note: Women not of childbearing potential are defined as: Any female who is post-menopausal [age > 55 years with cessation of menses for 12 or more months or less than 55 years but not spontaneous menses for at least 2 years or less than 55 years and spontaneous menses within the past 1 year, but currently amenorrheic (eg, spontaneous or secondary to hysterectomy), and with postmenopausal gonadotropin levels (luteinizing hormone and follicle-stimulating hormone levels > 40 IU/L) or postmenopausal estradiol levels (< 5 ng/dL) or according to the definition of "postmenopausal range" for the laboratory involved] or who have had a hysterectomy, bilateral salpingectomy, or bilateral oophorectomy). 25 | Page Version 6-26-2018
18. Sexually active subjects and their partners unwilling to use male latex condom to avoid potential viral transmission during sexual contact while on treatment and within 30 days after treatment with talimogene laherparepvec.
19. Subject who is unwilling to minimize exposure with his/her blood or other body fluids to individuals who are at higher risks for HSV-1 induced complications such as immunosuppressed individuals, individuals known to have HIV infection, pregnant women, or children under the age of 1 year, during talimogene laherparepvec treatment and through 30 days after the last dose of talimogene laherparepvec.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2018-12-20 (Actual); Primary Completion 2023-07-19 (Actual); Study Completion 2023-07-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clara Curiel, MD, Principal Investigator — University of Arizona
Locations (2):
- United States (2):
  - Honor Health Research Institute, Scottsdale, Arizona
  - University of Arizona Cancer Center, Tucson, Arizona

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: Target Injected Lesions
Groups:
- Treatment (Talimogene Laherparepvec): The subject participation period was approximately 48 weeks. This included a screening visit, 4 injection visits and 5 follow up visits. Total length of study/patient was 8.5 to 10.5 months. TVEC was administered by injection with a needle directly into one or more tumors.
Period: Overall Study
Arm/Group | Treatment (Talimogene Laherparepvec)
Started | 11; 24 Target Injected Lesions
Completed | 11; 24 Target Injected Lesions
Not Completed | 0; 0 Target Injected Lesions

BASELINE CHARACTERISTICS:
Units Other Than Participants: Target Injected Lesions
Arm/Group | Treatment (Talimogene Laherparepvec)
Number analyzed (Participants) | 11
Number analyzed (Target Injected Lesions) | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 0
  >=65 years | 11
Age, Continuous [Mean (Standard Deviation); unit: Years] | 75.7 (6.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 11
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 11
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 11
Number of TILs per participant [Count of Participants; unit: Participants] — The number of participants with 1, 2, or 4 target injected lesions (TILs)
  Participants
    1 TIL | 4
    2 TILs | 4
    4 TILs | 3
Tumor subtype of TILs [Count of Units; unit: Target Injected Lesions] — The number of individual TILs with keratoacanthoma or non-keratoacanthoma tumor subtypes across the 11 patients enrolled on the trial.
  Target Injected Lesions
    Keratoacanthoma | 3
    Non-keratoacanthoma | 21

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate
Description: The primary end point is to evaluate the overall response rate (ORR) defined as proportion of subjects who achieved complete response (CR) and partial response (PR) in the cSCC Target injected lesions (TILs).
Time Frame: 8.5-10.5 months
Population: All participants who received at least one dose of treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Talimogene Laherparepvec)
Number analyzed (Participants) | 11
Participants
  Overall Response Rate (ORR) | 11
  Partial Response (PR) | 1
  Complete Response (CR) | 10
Statistical Analysis 1: Comparison: Treatment (Talimogene Laherparepvec); Test type: Other; p = 0.0005, One-sample binomial test; One-sample binomial test versus null hypothesis value of 0.50; Overall Response Rate = 100, 95% CI 1-sided [lower limit 76.2]

2. Secondary Outcome: Number of Participants With Events Requiring the Discontinuation of Study Drug
Description: 1. Number of participants with events requiring the discontinuation of study drug
  1. 75% or greater number of Target injection lesions (TILs) meeting criteria for withdrawal.
  2. Identification of high-risk features in one or more TILs during study participation.
  3. Persistent discomfort (consecutive weeks of lesion pain, burning, or itching of Grade 2 or more).
Time Frame: 8.5-10.5 months
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Talimogene Laherparepvec)
Number analyzed (Participants) | 11
Participants
  TILs meeting criteria for withdrawal | 0
  Identification of high-risk features | 0
  Persistent discomfort | 0

3. Secondary Outcome: Time of Response.
Description: To measure time of response in cSCC individual TILs.
Time Frame: 8.5-10.5 months
Population: All TILs across 11 patients enrolled on the trial that received at least one dose of treatment (24 TILs total).
Measure: Mean (Standard Deviation); unit: Days
Units Other Than Participants: Target Injected Lesions
Arm/Group | Treatment (Talimogene Laherparepvec)
Number analyzed (Participants) | 11
Number analyzed (Target Injected Lesions) | 24
Days | 48.7 (29.2)
Statistical Analysis 1: Comparison: Treatment (Talimogene Laherparepvec); Test type: Other — Descriptive statistics; Mean = 48.7, Standard Deviation 29.2

4. Secondary Outcome: Duration of Overall Response.
Description: To measure the duration of overall response (DOR) of individual TILs.
Time Frame: 8.5-10.5 months
Population: All TILs across 11 patients enrolled on the trial that received at least one dose of treatment (24 TILs total).
Measure: Mean (Standard Deviation); unit: Days
Units Other Than Participants: Target Injected Lesions
Arm/Group | Treatment (Talimogene Laherparepvec)
Number analyzed (Participants) | 11
Number analyzed (Target Injected Lesions) | 24
Days | 201.4 (29.6)

5. Secondary Outcome: Assess Durable Response.
Description: Assess durable response rate (DRR) of TILs. DRR was assessed when the time of CR or PR with response lasting continuously for at least 6 months.
Time Frame: 8.5-10.5 months
Population: All TILs across 11 patients enrolled on the trial that received at least one dose of treatment (24 TILs total).
Measure: Number; unit: Percentage of individual TILs with DRR
Units Other Than Participants: Target Injected Lesions
Arm/Group | Treatment (Talimogene Laherparepvec)
Number analyzed (Participants) | 11
Number analyzed (Target Injected Lesions) | 24
Percentage of individual TILs with DRR | 83.3
Statistical Analysis 1: Comparison: Treatment (Talimogene Laherparepvec); Test type: Other — Binomial proportion of TILs; Percentage = 83.3

6. Secondary Outcome: Time to Progression.
Description: To measure the time to progression (TTP) of individual TILs.
Time Frame: 8.5-10.5 months
Population: All TILs across 11 patients enrolled on the trial that received at least one dose of treatment (24 TILs total).
Measure: Number; unit: Days
Units Other Than Participants: Target Injected Lesions
Arm/Group | Treatment (Talimogene Laherparepvec)
Number analyzed (Participants) | 11
Number analyzed (Target Injected Lesions) | 24
Days | NA — No TILs progressed.

7. Secondary Outcome: Overall Response Rate by Ultrasound.
Description: Overall response rate (ORR) (CR+PR) assessed by imaging technique (high frequency ultrasound). The subjects received ultrasound assessments of their TILs at baseline/screening visit (0), and at visit 6 (first follow up visit, approximately 4-5 months from baseline).The tumor volume change was assessed between the 2 visits, and percent of subjects with tumor volume reduction was reported.
Time Frame: Baseline and 4-5 months
Population: The barriers for collecting this data in clinic was both due to the COVID-19 pandemic and limited staffing at the lead institution's imaging department.
Measure: Number; unit: Percentage of participants
Arm/Group | Treatment (Talimogene Laherparepvec)
Number analyzed (Participants) | 5
Percentage of participants | 60

8. Secondary Outcome: Overall Clinical Response Rate - Targeted Lesions.
Description: Overall clinical response rate (CR+PR) of individual TILs with talimogene laherparepvec (not as overall subject response).
Time Frame: 8.5-10.5 months
Population: All TILs across 11 patients enrolled on the trial that received at least one dose of treatment (24 TILs total).
Measure: Number; unit: Count of TILs
Units Other Than Participants: Target Injected Lesions
Arm/Group | Treatment (Talimogene Laherparepvec)
Number analyzed (Participants) | 11
Number analyzed (Target Injected Lesions) | 24
Count of TILs
  ORR of individual TILs | 24
  PR of individual TILs | 1
  CR of individual TILs | 23
Statistical Analysis 1: Comparison: Treatment (Talimogene Laherparepvec); Test type: Other — Counts of TILs; Percentage = 100

9. Secondary Outcome: Percentage of Participants With Overall Clinical Response Rate - Non-injected Lesion(s).
Description: Percentage of Participants with overall clinical response rate (CR+PR) in cSCC Target non-injected lesion(s) (TNILs).
Time Frame: 8.5-10.5 months
Population: Target, non-injected lesions of participants who received at least one dose of treatment in a TIL. Only 2 participants had non-injected lesions and received at least one dose of treatment in a TIL.
Measure: Number; unit: Percentage of participants
Arm/Group | Treatment (Talimogene Laherparepvec)
Number analyzed (Participants) | 2
Percentage of participants | 100
Statistical Analysis 1: Comparison: Treatment (Talimogene Laherparepvec); Test type: Other; Percentage = 100

10. Secondary Outcome: Number of Safety Adverse Events (SAE) as Assessed According to the NCI Common Terminology Criteria for Adverse Events (CTCAE) 4.0
Description: 1. Number of safety adverse events (SAE) as assessed according to the NCI Common Terminology Criteria for Adverse Events (CTCAE) 4.0
  a. Clinically significant laboratory values i. Clinically significant laboratory values are based on participant condition and side effect. These will vary and will be determined by the clinical judgement of the research healthcare provider. Note: laboratory values will be collected for initial participant screening and side effects only, no other clinical laboratory values are scheduled in this protocol.
Time Frame: 8.5-10.5 months
Measure: Number; unit: Number of safety adverse events assessed
Arm/Group | Treatment (Talimogene Laherparepvec)
Number analyzed (Participants) | 11
Number of safety adverse events assessed | 21

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were assessed and collected starting from the first study treatment visit and continued through the last study follow-up visit, up to 10.5 months
Arm/Group | Treatment (Talimogene Laherparepvec)
All-Cause Mortality (participants affected / at risk) | 0/11
Serious Adverse Events (participants affected / at risk) | 0/11
Other Adverse Events (participants affected / at risk) | 9/11
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Talimogene Laherparepvec) (N=11)
Fatigue (General disorders) | 5 (11)
Flu-like symptoms (General disorders) | 4 (10)
Headache (Nervous system disorders) | 2 (5)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Chills (General disorders) | 1 (2)
Fever (General disorders) | 1 (1)
Injection site pain (General disorders) | 1 (1)
Leg pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Malaise (General disorders) | 1 (4)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (4)
Paresthesia (Nervous system disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-07-24): https://cdn.clinicaltrials.gov/large-docs/28/NCT03714828/Prot_SAP_000.pdf
  • Informed Consent Form (2022-12-22): https://cdn.clinicaltrials.gov/large-docs/28/NCT03714828/ICF_001.pdf